CLINICAL TRIAL: NCT07325162
Title: Development of a Next-Generation Optical Biometer for Eyes With Cataract
Brief Title: Development of Optical Biometer
Acronym: CH-0203
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cassini Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0203
Record Dates: First submitted 2025-12-04; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cataract and IOL Surgery
Keywords: Optical Biometer; SS-OCT
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All enrolled subjects (Other): All eligible subjects will undergo ocular biometry using three devices:
  1. the investigational optical biometer,
  2. Comparator Device A, and
  3. Comparator Device B. Measurements from all devices will be obtained at the same visit and used only for diagnostic comparison. No treatment assignment occurs.
  Interventions: Device: New Investigational Optical Biometer (Device); Device: Comparator Device A (Cassini Ambient); Device: omparator Device B (Argos)

INTERVENTIONS:
Device: New Investigational Optical Biometer (Device) — Investigational optical biometer used to obtain axial length, keratometry, anterior chamber depth, lens thickness, and total corneal astigmatism. Device is being evaluated for measurement accuracy and agreement.
Device: Comparator Device A (Cassini Ambient) — FDA-cleared corneal topographer used as a reference standard comparator for keratometry.
Device: omparator Device B (Argos) — FDA-cleared optical biometer used as a second comparator to assess agreement and measurement differences.

SUMMARY:
The Helioscope (Cassini Technologies B.V.) is a novel device under development that aims at combining LED-based corneal topography and SS-OCT to provide accurate and fast measurements of both the corneal shape and the ocular biometry. To that end, the hardware and software of the Cassini color-LED topographer (Cassini Technologies B.V.) is combined with a novel SS-OCT device.

While the new Helioscope can largely be evaluated using data acquired with healthy eyes, one of its main use-cases is providing input for IOL power formulae for cataract surgery. Thus, it is essential that the device can perform measurements in eyes with (dense) cataract. As cataract changes the optical properties of the crystalline lens and the OCT measurement is optical, this is not a given. This study therefore seeks a dataset of Helioscope measurements performed in eyes with cataract that can be used to develop the software algorithms of the Helioscope.

ELIGIBILITY:
Inclusion criteria:

* The presence of cataract in at least one eye.
* Minimally 21 years of age.
* Provided written informed consent.

Exclusion criteria:

* The inability to properly fixate on a fixation target for several seconds
* The inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Ocular parameters of cataractous eyes measured with a novel biometer | Overall study to complete up to 12 months
  Primary endpoint:
  Biometric ocular parameters of axial length, anterior chamber depth, central corneal thickness, keratometry, lens thickness and limbal white to white will be measured by the Helioscope device in 200 eyes.

SECONDARY OUTCOMES:
Comparison of ocular biometry measured by a novel biometer against FDA approved devices for planning cataract surgery | Overall study to complete up to 12 months
  Ocular biometric values (axial length, anterior chamber depth, keratometry, limbal white to white, lens thickness, and central corneal thickness - measured in millimetres) measured by the Helioscope device will be compared against the same values captured by the Argos biometer and Ambient topographer devices (both FDA approved devices on label use) in 200 eyes.

CONTACTS AND LOCATIONS:
Locations (1):
- Bishop Eye Center, Hilton Head Island, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because, although the data are randomized, they are being used to develop and validate proprietary software algorithms for the investigational device.

REFERENCES:
- [Result] Hashemi H, Sardari S, Yekta A, Khabazkhoob M. The repeatability and agreement of biometric measurements by dual Scheimpflug device with integrated optical biometer. Sci Rep. 2022 May 11;12(1):7748. doi: 10.1038/s41598-022-11953-8. PMID 35546610